CLINICAL TRIAL: NCT05742490
Title: Neonatal Infection Surveillance Database
Acronym: neonIN
Status: Recruiting | Type: Observational
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 05.0093
Record Dates: First submitted 2023-01-19; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: Neonatal Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NeonIN is a is a neonatal infection surveillance database which will facilitate active surveillance for bacterial infections through a network of neonatal units, using standardised definitions, proformas and microbiological techniques. The centralised and secure web-based database will allow real-time entry of data and rapid and timely analysis of results.

DETAILED DESCRIPTION:
The neonIN surveillance network captures data on episodes of invasive neonatal infection on a web-based database (www.neonin.org.uk). Over 25 UK neonatal units currently contribute to this database in real-time. An episode of neonatal infection is defined as a positive culture collected from a normally sterile site such as the blood, cerebrospinal fluid (CSF) or urine (via catheter or suprapubic aspirate) for which clinicians prescribed at least five days of appropriate antibiotics. Clinical, demographic and microbiological data (including antimicrobial susceptibilities) are collected using a standardised online questionnaire, and denominator data regarding the total number of live-births and neonatal-admissions are collected for each neonatal unit.

ELIGIBILITY:
Inclusion Criteria:

* Infants on participating Neonatal Units who have an episode of infection with a positive culture

Exclusion Criteria:

-

Ages: 1 Minute to 12 Months | Sex: All
Age Groups: Child
Study Population: Eligible infants will be identified from Neonatal Units
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2013-12-16 (Actual); Primary Completion 2023-11-22 (Estimated); Study Completion 2028-11-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of infection | 6 months
  Collection of neonIN data on episodes of significant neonatal bacterial infections in NNUs recruiting to neonIN
Antibiotic susceptibility | 6 months
  Collection of neonIN data on susceptibility profiles of significant neonatal bacterial infections
Features of bacterial infections | 6 months
  Collection of neonIN data on gestation, birth weight, age of onset, clinical presentation and prior antibiotic use of significant neonatal bacterial infections

CONTACTS AND LOCATIONS:
Overall Officials: Eva Galiza, MD, Principal Investigator — St George's, University of London
Locations (1):
- St George's University of London, London, United Kingdom

REFERENCES:
- [Background] Gkentzi D, Kortsalioudaki C, Cailes BC, Zaoutis T, Kopsidas J, Tsolia M, Spyridis N, Siahanidou S, Sarafidis K, Heath PT, Dimitriou G; Neonatal Infection Surveillance Network in Greece. Epidemiology of infections and antimicrobial use in Greek Neonatal Units. Arch Dis Child Fetal Neonatal Ed. 2019 May;104(3):F293-F297. doi: 10.1136/archdischild-2018-315024. Epub 2018 Jun 28. PMID 29954881
- [Background] Wang J, Kortsalioudaki C, Heath PT, Buttery J, Clarke P, Gkentzi D, Anthony M, Tan K; neonIN network. Epidemiology and healthcare factors associated with neonatal enterococcal infections. Arch Dis Child Fetal Neonatal Ed. 2019 Sep;104(5):F480-F485. doi: 10.1136/archdischild-2018-315387. Epub 2018 Nov 13. PMID 30425112
- [Background] Cailes B, Kortsalioudaki C, Buttery J, Pattnayak S, Greenough A, Matthes J, Bedford Russell A, Kennea N, Heath PT; neonIN network. Antimicrobial resistance in UK neonatal units: neonIN infection surveillance network. Arch Dis Child Fetal Neonatal Ed. 2018 Sep;103(5):F474-F478. doi: 10.1136/archdischild-2017-313238. Epub 2017 Oct 26. PMID 29074716
- [Background] Cailes B, Kortsalioudaki C, Buttery J, Pattnayak S, Greenough A, Matthes J, Bedford Russell A, Kennea N, Heath PT; neonIN network. Epidemiology of UK neonatal infections: the neonIN infection surveillance network. Arch Dis Child Fetal Neonatal Ed. 2018 Nov;103(6):F547-F553. doi: 10.1136/archdischild-2017-313203. Epub 2017 Dec 5. PMID 29208666
- [Background] Sapuan S, Kortsalioudaki C, Anthony M, Chang J, Embleton ND, Geethanath RM, Gray J, Greenough A, Lal MK, Luck S, Pattnayak S, Reynolds P, Russell AB, Scorrer T, Turner M, Heath PT, Vergnano S. Neonatal listeriosis in the UK 2004-2014. J Infect. 2017 Mar;74(3):236-242. doi: 10.1016/j.jinf.2016.11.007. Epub 2016 Nov 17. PMID 27867063